CLINICAL TRIAL: NCT06896422
Title: Prospective, Randomized Controlled Clinical Trial of Glutathione Combined With PD-1 Antibody and Chemotherapy in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Randomized Trial of Glutathione With Anti-PD-1 and Chemotherapy in Advanced NSCLC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yi Zhang, Director, Biotherapy Center, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-KY-0017-002
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-02

CONDITIONS: Non-Small Cell Lung Cancer; Chemotherapy; PD1 Antibody; Glutathione
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Glutathione; Immune Checkpoint Inhibitors; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PD-1 inhibitor plus chemotherapy arm (Placebo Comparator)
  Interventions: Drug: PD1 Inhibitor; Drug: Chemotherapy
- Glutathione combined with PD-1 inhibitor plus chemotherapy arm (Experimental)
  Interventions: Drug: Glutathione; Drug: PD1 Inhibitor; Drug: Chemotherapy

INTERVENTIONS:
Drug: Glutathione — Glutathione is administered as an adjunct intervention to the PD-1 inhibitor plus chemotherapy regimen.
  Arms: Glutathione combined with PD-1 inhibitor plus chemotherapy arm
Drug: PD1 Inhibitor — e.g. pembrolizumab, camrelizumab, sintilimab, tislelizumab, toripalimab
Drug: Chemotherapy — Platinum-based doublet chemotherapy

SUMMARY:
Chemotherapeutic agents exert significant immunomodulatory effects by influencing tumor-infiltrating immune cells. However, the sequence and combination of chemotherapy regimens differentially modulate immune cell dynamics, ultimately impacting treatment efficacy and patient survival. Glutathione, a critical bioactive molecule, demonstrates broad potential in tumor immunotherapy. Through mechanisms such as scavenging free radicals, modulating immune cell proliferation and differentiation, and regulating cytokine expression, glutathione achieves precise modulation of immune responses to enhance immune system functionality. To investigate whether glutathione can enhance the clinical efficacy of current chemo-immunotherapy regimens in non-small cell lung cancer (NSCLC), investigators conducted this clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of lung squamous cell carcinoma or adenocarcinoma.
2. Documented disease progression following first-line chemotherapy or chemo-immunotherapy.
3. Age ≥18 years at the time of enrollment.

Exclusion Criteria:

1. Patients with small cell lung cancer or other histological subtypes of lung cancer.
2. Patients lost to follow-up, who discontinued treatment, or died within one year of diagnosis.
3. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From randomization until the first documented disease progression or death from any cause, whichever occurs first, assessed up to 24 months."
Overall Response Rate (ORR) | From the initiation of treatment until 12 weeks
  Proportion of patients achieving predefined tumor volume reduction with sustained duration, defined as those attaining a complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Improvement in Immune Parameters | From baseline until 12 weeks post-treatment completion
  assess every 4 weeks via flow cytometry for peripheral CD8+ T-cell proportion and cytokine levels (e.g., IFN-γ, IL-2).
QLQ-LC43 | From baseline until 24 weeks post-treatment completion
  Quality of Life Questionnaire for Lung Cancer from the European Organization for Research and Treatment of Cancer (EORTC), assessed at baseline, the end of each treatment cycle (every 3 weeks), and at 12 and 24 weeks post-treatment using the Chinese version of the EORTC QLQ-LC43 questionnaire.
Overall survival | From randomization until death from any cause, assessed up to 60 months.
  the time from randomization (or treatment initiation) to death from any cause, serving as the gold-standard endpoint for evaluating long-term therapeutic efficacy in oncology.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No